CLINICAL TRIAL: NCT06792526
Title: Monitoring Salivary Gland Damage After Radiotherapy in Patients with Head and Neck Cancer Using Multimodal Radiomics
Brief Title: Prospective Study on Monitoring Parotid Gland Injury After Radiotherapy for Head and Neck Tumors Using Multimodal Radiomics
Status: Not yet recruiting | Type: Observational
Sponsor: Hainan People's Hospital (Other)
Responsible Party: Principal Investigator, Wu Wei, Principal Investigator (Graduate Research), Hainan People's Hospital
Other Study IDs: WuWei-2025-NPC002
Record Dates: First submitted 2025-01-12; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Xerostomia, Radiation-induced Parotid Damage,Predictivevalue,Head and Neck Cancer
MeSH Terms: conditions — Xerostomia; Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Head and Neck Cancer
  Interventions: Other: IVIM Imaging MRF Imaging

INTERVENTIONS:
Other: IVIM Imaging MRF Imaging — IVIM imaging will be performed to evaluate microstructural and perfusion changes in the salivary glands of Head and Neck Cancer undergoing radiotherapy. This technique quantifies diffusion and perfusion parameters, providing insights into early tissue damage. MRF imaging will be used to quantify salivary gland tissue characteristics, including relaxation parameters (T1 and T2 mapping), to monitor radiotherapy-induced damage. The technique enables precise tissue characterization through multi-parametric MRI.

SUMMARY:
Exploring a non-invasive and objective method for ultra early quantitative assessment of radiation-induced parotid gland injury. To provide a new and early method for evaluating changes in parotid gland function in clinical practice, and to guide the timing of interventions to protect the parotid gland.

DETAILED DESCRIPTION:
Exploring the application value of magnetic resonance fingerprinting (MRF) and intravoxel incoherent motion (IVIM) techniques in dynamically monitoring parotid gland injury and predicting the risk of dry mouth after radiotherapy for head and neck tumors. The study evaluated the changes in parotid gland cell density and microcirculation function by quantifying MRF (T1/T2 relaxation time, proton density) and IVIM parameters (D value, D * value, f value), combined with parotid gland volume reduction rate, to establish an early risk model for predicting dry mouth syndrome and optimize parotid gland protection strategies.

ELIGIBILITY:
Exclusion Criteria:

1. Contraindications to MRI, such as metallic implants or claustrophobia.
2. Severe comorbid conditions, including significant renal or hepatic dysfunction.
3. Concurrent participation in another interventional clinical trial.
4. Pregnant or breastfeeding.
5. Any condition that may impair compliance with study procedures.

Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of nasopharyngeal carcinoma.
2. Scheduled to undergo radiotherapy as part of standard treatment.
3. Aged 18 years or older.
4. No contraindications to MRI scans (e.g., no implanted metallic devices).
5. Written informed consent has been provided.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients (18 years of age or older) who have been diagnosed with a head and neck tumour and are planning to receive radiotherapy as part of their standard treatment. Recruitment will take place at the Department of Radiotherapy, Hainan Provincial People's Hospital. Applicants must be able to undergo an MRI scan and provide informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-01-20 (Estimated); Primary Completion 2025-07-20 (Estimated); Study Completion 2025-08-20 (Estimated)

PRIMARY OUTCOMES:
Quantitative assessment of salivary gland changes using IVIM and MRF imaging | From baseline to 3 months post-radiotherapy
  IVIM imaging will be performed to evaluate microstructural and perfusion changes in the salivary glands of Head and Neck Cancer undergoing radiotherapy. This technique quantifies diffusion and perfusion parameters, providing insights into early tissue damage. MRF imaging will be used to quantify salivary gland tissue characteristics, including relaxation parameters (T1 and T2 mapping), to monitor radiotherapy-induced damage. The technique enables precise tissue characterization through multi-parametric MRI.

IPD SHARING:
Plan to Share IPD: No